CLINICAL TRIAL: NCT06783634
Title: The Effect of High Single Dose of Dexamethasone in Prevention of Post-operative Acute Kidney Injury in Cardiac Surgeries Requiring Cardiopulmonary Bypass
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FMASU MS117/2024
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-02

CONDITIONS: Acute Kidney Injury After Adult Cardiac Surgery
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group : (Placebo Comparator): Group 1 (Control group) will receive normal saline as a placebo.
  Interventions: Drug: Placebo
- dexamethasone group (Active Comparator): Group 2 (dexamethasone group) single intra venous high dose of dexamethasone 1mg/kg with maximum dose of 100 mg.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Group 2 (dexamethasone group) single intra venous high dose of dexamethasone 1mg/kg with maximum dose of 100 mg.
  Arms: dexamethasone group
Drug: Placebo — Group 1 (Control group) will receive normal saline as a placebo.
  Arms: Control group :

SUMMARY:
The aim of the current study is to assess the effect of intra operative single high dose dexamethasone (1 mg/kg) in decreasing the incidence of post-operative acute kidney injury after cardiac surgeries with cardiopulmonary bypass

DETAILED DESCRIPTION:
Patients undergoing any type of elective cardiac surgical procedure requiring CPB will be randomly assigned into one of the following groups using computer generated codes (patients in each group):

* Group 1 (Control group) will receive normal saline as a placebo.
* Group 2 (dexamethasone group) single intra venous high dose of dexamethasone 1mg/kg with maximum dose of 100 mg.

  * Preoperative settings:

Preoperative assessment will be done to all the patients who were going to join this study before reaching the pre induction room.

The assessment will include:

* Full History taking.
* Full examination including the airway assessment. Checking the lab results (complete blood picture, prothrombin time, partial thromboplastin time, liver functions and viral markers and specially kidney function tests) and radiographic studies
* ECG and EChO

On reaching the pre-induction room, the following will be done for each patient included in the current study:

* Inserting a secured intravenous (I.V.) access in a sterile technique.
* Antibiotic will be given I.V. after sensitivity test is done.
* Anti-stress medication (e.g. lansoprazole 60 mg) will be given I.V. slowly diluted in a 20 ml normal saline to be repeated every 12 hours (Avner et al., 1995).
* Sedation will be given in the form of 1-2 mg of Midazolam.
* Attaching a monitor (pulse oximetry, non-invasive blood pressure, 5-lead ECG) till the patient enter the OR with recording the initial vital data.

  * Intraoperative settings:

After lying of the patient down on the OR table:

* Basic monitoring leads (5-lead ECG, pulse oximeter, invasive blood pressure IBP) will be attached to the patient with recording the basal vital data.
* I.V. crystalloid ringer solution will be started and maintained all through the operation.
* An arterial 20G vygon cannula will be inserted in the radial artery of the non-dominant hand, and connected to an arterial dome through a non-compliant A-line. Thus, obtaining arterial blood gas (ABG) samples during the operation, and continuous beat-to-beat blood pressure monitoring (Pierre et al., 2018).
* Pre-induction oxygenation with 100% oxygen will be done for 1 minute.
* Induction using an opioid-based general anesthesia will be done by giving 0.03 - 0.05 mg/kg of Midazolam (Midathetic® Amoun Pharm, a 5 mg/1 ml ampoule) (Lingamchetty et al., 2019), 1 mg/kg of Propofol (Propofol 1% Fresenius®, a 200 mg/20 ml ampoule) (Folino et al., 2022), 3-5 mcg/kg of Fentanyl (Fentanyl hameln® Sunny Pharmaceutical Company, a 100 mcg/2 ml ampoule) (Bailey et al., 1985), 0.5-0.6 mg/kg of Atracurium (Atrabesylate® EGY Pharm, a 50 mg/5 ml ampoule) (Chalermkitpanit et al., 2020), and supporting the patient's ventilation for 2-4 minutes.

Tracheal intubation will be performed by an experienced anesthesiologist. A lubricant will be used on the tip of the endotracheal tube (ETT) before intubation

* Mechanical ventilation will be controlled by adjusting the current volume to 8-10 mL/Kg and frequency of ventilation of up to 12-14 breaths/min to maintain normocapnia: end-tidal pressure CO2 (ET CO2) at the level of 35 ± 5 mm Hg and respiratory frequency, oxygen: air 50%: 50%
* An ultrasound-guided insertion of triple line 7 Fr. Central venous catheter (CVC) in the right/left internal jugular vein will be done after full sterilization with chlorhexidine with contact time 1-2 minutes and sterile draping to the site of insertion.
* A temperature probe will be applied to the patient
* Anesthesia is going to be maintained using isoflurane (1.0 - 1.5%), oxygen (1-2 lit/min) and air (1-2 lit/min), by means of a circuit with CO2 absorption. Neuromuscular blockage is going to be maintained by Atracurium infusion with a rate 0.3 mg/kg/hr. to guarantee that the patient was fully paralyzed all through the surgery.

Patients will be randomized to receive either dexamethasone or placebo treatment. Dexamethasone (1mg/kg of body weight, with a 100mg maximum) or placebo will be administered as a single intravenous injection after induction of anesthesia, but before initiation of CPB.

The study drug will be supplied in packaged ampoules, each assigned to a unique study number. Packages and ampoules of dexamethasone and placebo will be identical and contain an equal volume of either a dexamethasone (Dexamethasone - MUP 8 MG / 2 ML (Dexamethasone Sodium Phosphate) solution or normal saline, respectively. The research pharmacist, will prepare and deliver batches of (60) ampoules. When a consenting patient arrive in the operating department, a packaged ampoule will be taken from the batch.

When the ampoule is opened and the study drug is administered, the patient is considered randomized and the corresponding study number will be assigned to that patient. Patients, caregivers, and researchers will be unaware of study group assignment.

• Postoperative settings: After surgery, patients are transferred to the intensive care unit (ICU) and will be weaned from mechanical ventilation when there was no excessive ongoing blood loss and patients were cooperative and hemodynamically stable. Perioperative serum glucose is regulated according to local sliding scale protocols.

Post-operative serum creatinine, GFR will be obtained once daily, and hourly urine output will be followed for 7 days, acute kidney injury is defined according to the RIFLE criteria as an increase in postoperative serum creatinine of at least 2 to 3 times the preoperative baseline value or GFR decreased >25%, or urine output < 0.5 mL/kg/h >12 h, and failure defined as a serum creatinine level of more than 4 mg/dL associated with an acute increase of serum creatinine of at least 0.5 mg/dL (Bellomo et al., 2004).

Other measurements will be included as a secondary outcome as: the time used to wean of ventilator, the duration of ICU stay and duration till discharge from hospital, incidence of developing post-operative infection, glucose level will be obtained hourly for the first 24 hours then every 4 hours till ICU discharge then twice daily till completion of the 7 days of the study, the incidence of developing diabetic ketoacidosis (DKA) or hyperglycemic hyperosmolar coma also will be followed up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-65 years.
2. Sex: Both sex.
3. Patients with American Society of Anesthesiologists (ASA) score III - IV.
4. Patients who were scheduled for any type of elective cardiac surgical procedure requiring cardiopulmonary bypass

Exclusion Criteria:

1. Declining to give written informed consent.
2. History of allergy to the medications used in the study.
3. Emergent or planned off-pump procedure
4. Diabetic patients.
5. Patients with recent history of AKI, or have any renal deterioration as GFR < 80 ml/min./1.73/m2
6. Patients scheduled for urgent cardiac surgery.
7. Patients scheduled for ascending aortic surgery inducing deep hypothermic total circulatory arrest.
8. Patients on high doses of inotropes and/or vasopressors.
9. Patients with high drain(s) in the first 6 hours postoperatively.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-03-25 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
postoperative acute kidney injury | 7 days
  Measure the incidence of occurrence of postoperative acute kidney injury in each group of the patients included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Nourhan E Abdellatif, MBBCH, Principal Investigator — Anesthesia resident Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared once study is completed
Supporting Information: Study Protocol